CLINICAL TRIAL: NCT04484259
Title: Pharmacodynamic Effects of Different Ticagrelor Maintenance Dosing Regimens With and Without Aspirin in Patients With Diabetes Mellitus: The OPTIMUS (Optimizing Antiplatelet Therapy in Diabetes Mellitus)-7 Study
Brief Title: Ticagrelor With and Without Aspirin in Patients With Diabetes Mellitus
Acronym: OPTIMUS-7
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB202001694
Record Dates: First submitted 2020-07-21; First posted 2020-07-23 (Actual); Results first posted 2025-03-30 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Diabetes Mellitus, Type 2; Coronary Artery Disease
Keywords: diabetes mellitus; ticagrelor; clopidogrel; percutaneous coronary intervention
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Coronary Artery Disease; Diabetes Mellitus | interventions — Ticagrelor; Aspirin; Clopidogrel

STUDY DESIGN:
Intervention Model Description: Prospective randomized
Masking Description: Staff performing PK/PD assessments will remain blinded to treatment assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Ticagrelor (Experimental): ticagrelor 60 mg bid monotherapy
  Interventions: Drug: Ticagrelor monotherapy
- Aspirin plus Clopidogrel (Active Comparator): aspirin 81 mg qd plus clopidogrel 75 mg qd
  Interventions: Drug: Clopidogrel with aspirin
- Aspirin plus Ticagrelor (Active Comparator): aspirin 81 mg qd plus ticagrelor 60 mg bid
  Interventions: Drug: Ticagrelor plus aspirin

INTERVENTIONS:
Drug: Ticagrelor monotherapy — Eligible patients will enter a 7-10 day run-in phase with aspirin 81 mg/ qd plus ticagrelor 90 mg bid after which they will discontinue aspirin and maintain ticagrelor 90 mg bid monotherapy for 10±3 days. After this period, patients will be randomized using a randomly generated computer sequence in a 1:1:1 fashion to either: a) ticagrelor 60 mg bid monotherapy; b) aspirin 81 mg qd plus ticagrelor 60 mg bid; c) aspirin 81 mg qd plus clopidogrel 75 mg qd. Randomized treatment will be maintained for 10±3 days.
  Other Names: Brilinta
  Arms: Ticagrelor
Drug: Ticagrelor plus aspirin — Eligible patients will enter a 7-10 day run-in phase with aspirin 81 mg/ qd plus ticagrelor 90 mg bid after which they will discontinue aspirin and maintain ticagrelor 90 mg bid monotherapy for 10±3 days. After this period, patients will be randomized using a randomly generated computer sequence in a 1:1:1 fashion to either: a) ticagrelor 60 mg bid monotherapy; b) aspirin 81 mg qd plus ticagrelor 60 mg bid; c) aspirin 81 mg qd plus clopidogrel 75 mg qd. Randomized treatment will be maintained for 10±3 days.
  Other Names: Brilinta
  Arms: Aspirin plus Ticagrelor
Drug: Clopidogrel with aspirin — Eligible patients will enter a 7-10 day run-in phase with aspirin 81 mg/ qd plus ticagrelor 90 mg bid after which they will discontinue aspirin and maintain ticagrelor 90 mg bid monotherapy for 10±3 days. After this period, patients will be randomized using a randomly generated computer sequence in a 1:1:1 fashion to either: a) ticagrelor 60 mg bid monotherapy; b) aspirin 81 mg qd plus ticagrelor 60 mg bid; c) aspirin 81 mg qd plus clopidogrel 75 mg qd. Randomized treatment will be maintained for 10±3 days.
  Other Names: Plavix
  Arms: Aspirin plus Clopidogrel

SUMMARY:
Recent studies have shown that withdrawing aspirin and maintaining P2Y12 inhibitor monotherapy for up to 12 months post-PCI, after a brief period of DAPT, reduces bleeding without increasing ischemic harm. Such effects have shown to of particular benefit in patients with diabetes mellitus (DM). However, if an aspirin-free approach can be considered after this time frame is a matter of debate. The aim of this study is to assess the PD effects of ticagrelor 60 mg with and without aspirin therapy in CAD patients and to compare this with a standard DAPT regimen of aspirin plus clopidogrel.

DETAILED DESCRIPTION:
Dual antiplatelet therapy (DAPT) with aspirin and a P2Y12 inhibitor is the standard of care for the prevention of thrombotic complications in patients with coronary artery disease (CAD) undergoing percutaneous coronary interventions (PCI). However, such ischemic benefit occurs at the expense of enhanced bleeding, the risk of which increases in a graded fashion with prolonged exposure to DAPT. Recent studies have shown that withdrawing aspirin and maintaining P2Y12 inhibitor monotherapy for up to 12 months post-PCI, after a brief period of DAPT, reduces bleeding without increasing ischemic harm. Such effects have shown to of particular benefit in patients with diabetes mellitus (DM). However, if an aspirin-free approach can be considered after this time frame is a matter of debate. In fact, current guidelines recommend maintaining P2Y12 inhibiting therapy for high risk patients but which all imply background use of aspirin. P2Y12 inhibitors for long-term (beyond 12 months) secondary prevention mainly include clopidogrel and ticagrelor. In particular, the dosing regimen for clopidogrel remains the standard 75 mg qd, whereas ticagrelor dosing is recommended to be reduced from 90 mg bid to 60 mg bid. However, of these regimens the pharmacodynamics (PD) effects of ticagrelor 60 mg in the absence of aspirin has not yet been tested. Because DM patients are likely to continue with long-term P2Y12 inhibitor therapy, defining the optimal antithrombotic approach for these patients is of critical importance. In light of the above made observations, patients with DM represent an ideal population to define the antiplatelet effects of a ticagrelor 60 mg monotherapy regimen. The aim of this study is to assess the PD effects of ticagrelor 60 mg with and without aspirin therapy in CAD patients and to compare this with a standard DAPT regimen of aspirin plus clopidogrel.

ELIGIBILITY:
Inclusion criteria:

For inclusion in the study patients should fulfill the following criteria:

1. Provision of informed consent prior to any study specific procedures
2. Men or women ≥18 years of age
3. Diagnosed with type 2 DM defined by ongoing glucose lowering therapy (oral medications and/or insulin) treatment for at least 1 month
4. Known angiographically defined CAD (including a history of previous PCI, CABG, or >50% stenosis in a major epicardial vessel) on standard of care antiplatelet therapy* *Patients can be treated with any background antiplatelet treatment regimen as part of their standard of care, including aspirin and/or any P2Y12 inhibitor (clopidogrel, ticagrelor, prasugrel).

Exclusion criteria:

1. PCI < 6 months prior
2. Recent (< 6 months) type I myocardial infarction
3. Anticipated concomitant oral or intravenous therapy with strong cytochrome P450 3A4 (CYP3A4) inhibitors or CYP3A4 substrates with narrow therapeutic indices that cannot be stopped for the course of the study:

   * Strong inhibitors: ketoconazole, itraconazole, voriconazole, telithromycin, clarithromycin (but not erythromycin or azithromycin), nefazadone, ritonavir, saquinavir, nelfinavir, indinavir, atanazavir
   * CYP3A4 substrates with narrow therapeutic index: quinidine, simvastatin at doses >40 mg daily or lovastatin at doses >40 mg daily
4. Anticipated concomitant oral or intravenous therapry of strong CYP3A inducers (phenytoin, rifampin, phenobarb, carbamazepine)
5. Need for chronic oral anticoagulant therapy or chronic low-molecular-weight heparin (at venous thrombosis treatment not prophylaxis doses)
6. Patients with known bleeding diathesis or coagulation disorder
7. History of previous intracerebral bleed at any time, gastrointestinal (GI) bleed within the past 6 months prior to randomization, or major surgery within 30 days prior to randomization
8. Active pathological bleeding
9. Hypersensitivity to aspirin, ticagrelor or clopidogrel
10. Increased risk of bradycardic events (eg, known sick sinus syndrome, second or third degree AV block or previous documented syncope suspected to be due to bradycardia) unless treated with a pacemaker
11. Known severe liver disease
12. Renal failure requiring dialysis
13. Known platelet count <80x106/mL
14. Known hemoglobin <9 g/dL
15. Pregnant or breastfeeding women. *Women of childbearing age must use reliable birth control (i.e. oral contraceptives) while participating in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2021-03-31 (Actual); Primary Completion 2024-01-29 (Actual); Study Completion 2024-06-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dominick J Angiolillo, MD,PhD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 105 patients consented.
  * 4 screen failures
  * 16 withdrawn during run in
  * 4 lost to follow-up before randomization visit
Groups:
- Aspirin Plus Ticagrelor 90 mg: Eligible patients entered a 7-10 day run-in phase with aspirin 81 mg qd plus ticagrelor 90 mg bid
- Ticagrelor 90 mg Monotherapy: Patients discontinued aspirin and maintained ticagrelor 90 mg bid monotherapy for 10±3 days.
Period: Run-in Phase With Aspirin and Ticagrelor
Arm/Group | Ticagrelor | Aspirin Plus Clopidogrel | Aspirin Plus Ticagrelor | Aspirin Plus Ticagrelor 90 mg | Ticagrelor 90 mg Monotherapy
Started | 0 | 0 | 0 | 101 | 0
Completed | 0 | 0 | 0 | 82 | 0
Not Completed | 0 | 0 | 0 | 19 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 9 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 4 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 2 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 4 | 0
Period: Run-in Phase With Ticagrelor Monotherapy
Arm/Group | Ticagrelor | Aspirin Plus Clopidogrel | Aspirin Plus Ticagrelor | Aspirin Plus Ticagrelor 90 mg | Ticagrelor 90 mg Monotherapy
Started | 0 | 0 | 0 | 0 | 82
Completed | 0 | 0 | 0 | 0 | 81
Not Completed | 0 | 0 | 0 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 1
Period: Randomized Treatment
Arm/Group | Ticagrelor | Aspirin Plus Clopidogrel | Aspirin Plus Ticagrelor | Aspirin Plus Ticagrelor 90 mg | Ticagrelor 90 mg Monotherapy
Started | 26 | 27 | 28 | 0 | 0
Completed | 25 | 27 | 28 | 0 | 0
Not Completed | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ticagrelor | Aspirin Plus Clopidogrel | Aspirin Plus Ticagrelor | Total
Number analyzed (Participants) | 26 | 27 | 28 | 81
Age, Continuous [Mean (Standard Deviation); unit: years] | 63 (8) | 65 (8) | 65 (10) | 64 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 7 | 13 | 36
  Male | 10 | 20 | 15 | 45
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 10 | 8 | 4 | 22
  White | 16 | 18 | 23 | 57
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 0 | 1
Hemoglobin A1c [Mean (Standard Deviation); unit: % of glycated hemoglobin] | 8.0 (2.0) | 7.5 (2.7) | 7.6 (2.4) | 7.7 (2.0)

OUTCOME MEASURES:

1. Primary Outcome: P2Y12 Reaction Units (PRU)
Description: The primary end-point of the study is the comparison of the PRU determined by VerifyNow PRU between between aspirin plus ticagrelor 60 mg and ticagrelor 60 mg monotherapy (trough effect pre-dosing). The VerifyNow System is a turbidimetric based optical detection system which measures platelet induced aggregation as an increase in light transmittance. The assay is based on microbead agglutination induced by adenosine diphosphate (ADP). The instrument measures this change in optical signal and reports results in P2Y12 Reaction Units (PRU).
Time Frame: Day 10, pre-dose
Measure: Mean (95% Confidence Interval); unit: PRU
Arm/Group | Ticagrelor | Aspirin Plus Clopidogrel | Aspirin Plus Ticagrelor
Number analyzed (Participants) | 26 | 27 | 28
PRU | 47 [26 to 68] | 136 [110 to 162] | 39 [20 to 57]
Statistical Analysis 1: Comparison: Ticagrelor; The primary end point was non-inferiority of Ticagrelor 60 mg monotherapy vs. aspirin plus Ticagrelor 60 mg; Test type: Non-Inferiority — non-inferiority margin 45 PRU; Mean Difference (Final Values) = 7, 95% CI 2-sided [-23 to 38]

2. Other Pre Specified Outcome: VASP
Description: Comparison of the platelet reactivity index (PRI) determined by VASP between between aspirin plus ticagrelor 60 mg and ticagrelor 60 mg monotherapy. VASP phosphorylation (VASP-P) is a marker of P2Y12 receptor signaling. VASP was assessed the ELISA VASP-P kit. Low PRI indicates appropriate platelet inhibition.
Time Frame: Day 10, pre-dose
Measure: Mean (95% Confidence Interval); unit: PRI
Arm/Group | Ticagrelor | Aspirin Plus Clopidogrel | Aspirin Plus Ticagrelor
Number analyzed (Participants) | 26 | 27 | 28
PRI | 77 [72 to 82] | 73 [68 to 78] | 70 [66 to 76]

3. Other Pre Specified Outcome: Comparison of Platelet Aggregation With ADP as Stimuli Determined by Light Transmittance Aggregometry Between Between Aspirin Plus Ticagrelor 60 mg and Ticagrelor 60 mg Monotherapy.
Description: Platelet aggregation was stimulated by ADP. Platelet aggregation will be determined as the maximal percent change (MPA%) in light transmittance from baseline. Low MPA% reflects good platelet inhibition.
Time Frame: Day 10, pre-dose
Measure: Mean (95% Confidence Interval); unit: MPA%
Arm/Group | Ticagrelor | Aspirin Plus Clopidogrel | Aspirin Plus Ticagrelor
Number analyzed (Participants) | 26 | 27 | 28
MPA% | 29 [23 to 36] | 39 [33 to 45] | 26 [20 to 32]

4. Other Pre Specified Outcome: Comparison of Thrombus Formation Measured by T-TAS Between Between Aspirin Plus Ticagrelor 60 mg and Ticagrelor 60 mg Monotherapy
Description: T-TAS is an automated microchip flow chamber system for the quantitative analysis of the thrombus formation process under blood flow conditions. In the present study, total platelet-derived thrombus formation is expressed as the area under the flow pressure curve for the first 10 min for the PL-chip tested at a flow rate of 18 μL/min (PL18-AUC10). Results of the assay are reported as PL18-AUC10. Low AUC reflect reduced thrombus growth and rapid breakdown of the thrombus.
Time Frame: Day 10, pre-dose
Measure: Mean (95% Confidence Interval); unit: kPa x minutes
Arm/Group | Ticagrelor | Aspirin Plus Clopidogrel | Aspirin Plus Ticagrelor
Number analyzed (Participants) | 26 | 27 | 28
kPa x minutes | 258 [207 to 308] | 147 [98 to 196] | 67 [19 to 115]

ADVERSE EVENTS:
Time Frame: 10 days
Description: These adverse event reporting reflects adverse events occurred during the randomized phase of the study.
Groups:
- Aspirin Plus Ticagrelor 90 mg: 7-10 day run-in phase with aspirin 81 mg qd plus ticagrelor 90 mg bid
- Ticagrelor 90 mg Monotherapy: discontinue aspirin and maintain ticagrelor 90 mg bid monotherapy for 10±3 days
Arm/Group | Ticagrelor | Aspirin Plus Clopidogrel | Aspirin Plus Ticagrelor | Aspirin Plus Ticagrelor 90 mg | Ticagrelor 90 mg Monotherapy
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/27 | 0/28 | 0/101 | 0/82
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/27 | 0/28 | 2/101 | 0/82
Other Adverse Events (participants affected / at risk) | 7/26 | 12/27 | 7/28 | 7/101 | 0/82
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ticagrelor (N=26) | Aspirin Plus Clopidogrel (N=27) | Aspirin Plus Ticagrelor (N=28) | Aspirin Plus Ticagrelor 90 mg (N=101) | Ticagrelor 90 mg Monotherapy (N=82)
iliac artery perforation (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Common iliac artery perforation and intra-abdominal bleeding occurred during a procedure that was performed per standard of care
chest pain (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ticagrelor (N=26) | Aspirin Plus Clopidogrel (N=27) | Aspirin Plus Ticagrelor (N=28) | Aspirin Plus Ticagrelor 90 mg (N=101) | Ticagrelor 90 mg Monotherapy (N=82)
dyspnea (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 12 (12) | 7 (7) | 7 (7) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-10-27): https://cdn.clinicaltrials.gov/large-docs/59/NCT04484259/Prot_SAP_000.pdf